CLINICAL TRIAL: NCT03026192
Title: Use of Near Infrared Spectroscopy in Preterm Infants to Determine Patent Ductus Arteriosus Closure Following Medical Treatment
Brief Title: Near Infrared Spectroscopy to Determine Patent Ductus Arteriosus Closure
Status: Terminated | Type: Observational
Why Stopped: not enough patients enrolled in study
Sponsor: Albany Medical College (Other)
Responsible Party: Principal Investigator, Kate Tauber, Assistant Professor, Albany Medical College
Other Study IDs: 4585
Record Dates: First submitted 2017-01-18; First posted 2017-01-20 (Estimated); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Patent Ductus Arteriosus
MeSH Terms: conditions — Ductus Arteriosus, Patent | interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- no PDA: These are infants who do not have a patent ductus arteriosus (PDA) as determine by echocardiography
  Interventions: Device: near infrared spectroscopy
- hsPDA: These are infants who have a hemodynamically significant PDA (hsPDA) as determined by echocardiography
  Interventions: Device: near infrared spectroscopy

INTERVENTIONS:
Device: near infrared spectroscopy — Near infrared spectroscopy will be placed on infants both with and without hsPDA

SUMMARY:
Using cerebral and renal near infrared spectroscopy monitoring to determine PDA closure in preterm infants after completing medical treatment for a hemodynamically significant PDA.

ELIGIBILITY:
Inclusion Criteria:

* preterm infants less than 32 weeks gestation

Exclusion Criteria:

* infection, congenital heart disease, syndromic anomalies, and perinatal asphyxia.

Ages: 1 Minute to 1 Week | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Preterm infants both with and without hsPDA. They will have NIRS monitors placed to measure cerebral and renal regional tissue oxygenation. Those without a hsPDA will be monitored solely around the time of initial echocardiogram. Those with a hsPDA will be monitored around initial echocardiogram and the subsequent echocardiogram after treatment completion.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2016-12; Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Change in NIRS readings | 3 days

CONTACTS AND LOCATIONS:
Locations (1):
- Albany Medical Center Neonatal Intesive Care Unit, Albany, New York, United States

IPD SHARING:
Plan to Share IPD: No